CLINICAL TRIAL: NCT05454696
Title: Effects of Online Clinic Pilates Exercises on Functionality and Physical Fitness in Patients Undergoing Bariatric Surgery
Brief Title: Online Clinic Pilates Exercises in Patients Undergoing Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Goksen Kuran Aslan, Associated Proffesor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/GAslan
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Bariatric Surgery; Obesity; Exercise; Physical Activity
Keywords: Physical Fitness; Exercise; Pilates; Quality of Life
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): The exercise group will follow the online clinical mat pilates exercises (via Zoom application) accompanied by a physiotherapist.
  Interventions: Other: Exercise
- Control Group (Active Comparator): The control group will receive online (via Zoom application) physical activity counselling by the physiotherapist only once.
  Interventions: Other: online physical activity counselling

INTERVENTIONS:
Other: Exercise — Patients in the exercise group will participate in online clinical pilates exercise sessions under the supervision of a physiotherapist twice a week. The exercises will be done via the Zoom application and will continue for 6 weeks. The exercise program will last one hour with a warm-up and cool-down period. The exercises will be done by adhering to the basic principles of clinical pilates. The exercise program includes mat exercises that provide general body strengthening and stretching. Progression will be provided according to the health status of the patients and their compliance with exercise. The intensity of exercise will be planned as medium according to the Rating of perceived exertion (RPE) Scale.
  Arms: Exercise Group
Other: online physical activity counselling — CG will receive online physical activity counselling by a physiotherapist only once. The importance of physical activity after surgery and the points to be considered during physical activity will be explained to the patients.
  Arms: Control Group

SUMMARY:
Obesity is defined as abnormal or excessive fat accumulation that can impair health. Obesity is considered a risk factor for diseases such as hypertension, heart failure, coronary heart diseases, diabetes mellitus, sleep apnea, and osteoarthritis. The prevalence of obesity is increasing all over the world. Therefore, it is very important to decide on the most appropriate treatment therapy method for the treatment of obesity. Bariatric surgery has become an accepted method in the treatment of obesity in recent years. It is the most effective and efficient treatment method in the long term for individuals with severe obesity. Exercise therapy is recommended by literature to maintain weight loss, prevent weight regain and minimize complications after bariatric surgery. However, there is no consensus on the appropriate exercise program. There is heterogeneity in the type, intensity and duration of exercise. In addition, the effect of clinical pilates exercises in the post-bariatric period has not been examined. Moreover, there is no study conducted in the post-bariatric period with telerehabilitation, which has been very popular in recent years. This study aims to reveal the effect of clinical pilates exercises on the functionality and physical fitness of post-bariatric patients. The results of our study will also contribute to the literature by revealing the effect of telerehabilitation on these patients.

DETAILED DESCRIPTION:
Patients who have undergone bariatric surgery and are followed in the Department of Endocrinology and Metabolism of Istanbul University Faculty of Medicine will be included in this study. Pre-treatment evaluation of the participants will be made and then individuals will be divided into two groups as Exercise Group (EG) and Control Group (CG) with a computer-assisted randomization program. The study will be conducted in accordance with the Declaration of Helsinki and a consent form will be obtained from the patients. Before the study, the purpose of the study will be explained and detailed information will be provided to the patients. CG will receive online physical activity counselling by a physiotherapist only once. EG will do online clinical pilates exercises under the supervision of a physiotherapist. The exercise program will last for 1 hour with a warm-up and cool-down period and the program will be continued twice a week for a total of 6 weeks. At the end of the treatment, individuals will be evaluated again. The primary aim is to examine the effect of online clinical pilates exercises on functionality and physical fitness in patients undergoing bariatric surgery. The secondary aim is to examine the effectiveness of telerehabilitation program after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 60
* Patients who volunteer
* Patients who can use technological devices at a level to participate in the online treatment
* Patients who completed a minimum of 8 weeks and a maximum of 2 years after surgery

Exclusion Criteria:

* Patients who are pregnant
* Patients who have psychiatric or psychological disorders that may affect adherence to treatment
* Patients who have an orthopaedic, neurological, cardiac, pulmonary or metabolic condition that may prevent participation and continuation of the exercise program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The Senior Fitness Test | 6 weeks
  The Senior Fitness Test Battery is used to evaluate the functional status of the participants. This battery consisted of 6 different tests that assess cardiorespiratory fitness, muscle strength, endurance and flexibility. Although it is a test that is developed to assess the functional evaluation of elderly individuals, it is used for functional evaluation of cases with fibromyalgia and obesity.
Six-Minute Walk Test (6 MWT) | 6 weeks
  The 6 MWT is used to evaluate the aerobic endurance of the patients. 6 MWT will be done according to American Thoracic Society (ATS) criteria. This test requires patients to walk at their own walking pace, as fast as possible but without running, for 6 minutes on a 30-metre straight corridor and the distance covered in meters will be recorded. In addition, before and after saturation, heart rate, dyspnea and fatigue levels will be evaluated by pulse oximetry. Modified Borg Dyspnea and Fatigue Scales will be used to determine dyspnea and fatigue levels.
The Chair Stand Test | 6 weeks
  This test is used to assess lower extremity strength and function. This requires participants to repeatedly stand up from and sit down on a chair for 30 seconds. The number of stands will be recorded.
The Biceps Curl Test | 6 weeks
  This requires participants to repeatedly lift a 5 lb (2.27 kg) weight (for women) or an 8 lb (3.63 kg) weight (for men) for 30 seconds. The number of lifts will be recorded. This reflects upper body strength.
The Chair Sit and Reach Test | 6 weeks
  For the test, the individual is asked to reach towards the toes with both hands in a sitting position with one knee flexed, the other knee extended and the ankle flexed to 90 degrees. The distance between the tip of the finger and the tip of the toe is recorded in cm. The test is repeated three times, the best distance is recorded, and the test is repeated for both limbs. This reflects lower body flexibility.
The Back Scratch Test | 6 weeks
  One hand is extended over the shoulder and the other is extended up the middle of the back and the approach distance of the middle fingers is measured and recorded in centimetres (cm). The test is repeated three times, the best distance is recorded, and the test is repeated for both limbs. This reflects upper body flexibility.
8-Foot Up and Go Test | 6 weeks
  This test requires the patient to get up from the chair as quickly as possible, take 8 steps and sit back in the chair. The time that's spent is measured and recorded in seconds.

SECONDARY OUTCOMES:
Muscle Strength | 6 weeks
  A digital dynamometer is used to evaluate muscle strength. Muscle strength is recorded in Newtons (N). Each measurement is repeated three times for the right and left extremities and the average recorded.
Core Stabilization | 6 weeks
  Core stability is evaluated with the Pressure Biofeedback Unit in accordance with the Sahrmann Core Stability Test protocol. The cuff is placed on the natural lordotic curve and inflated to 40 mmHg while the patient is lying supine. The test consists of 5 levels, while different lower extremity movements are performed at each level, core stabilization is expected to be preserved. After the patient completes a level successfully, other levels are tried.
Obesity and Weight Loss Quality Of Life (OWLQOL) | 6 weeks
  The Obesity and Weight Loss Quality of Life Scale, developed by Patrick et al., is used to assess the health-related quality of life of patients. The scale is single-factor and has no sub-groups. The scale consists of 17 items and each item is scored between 0-6. A single quality of life score is obtained by summing all of the items. The higher score is related to high quality of life.
Nottingham Health Profile | 6 weeks
  The Nottingham Health Profile (NHP) is a general patient-reported outcome measure which seeks to measure subjective health status. It is a questionnaire designed to measure a patient's view of their own health status in several areas. The NHP is consisted of two parts; the first part focuses on health and comprises 38 items which deal with pain, energy, sleep, mobility, emotional reaction and social isolation. The second part focuses on life areas affected and consists of 7 items which deal with problems regarding occupation, housework, social life, family life, sexual function, hobbies and holidays. The second part of the NHP is optional and can be omitted without ruining the test results.
Body Fat Percentage | 6 weeks
  The body fat percentage (BFP) of a patient is the total mass of fat divided by total body mass, multiplied by 100; body fat includes essential body fat and storage body fat. The body fat percentage of the patients will be evaluated with the bioelectrical impedance analysis technique. Results will be recorded in percent.
Muscle Mass | 6 weeks
  Muscle mass means the amount of soft muscle tissue in the body. The muscle mass of the patients will be evaluated with the bioelectrical impedance analysis technique. Results will be recorded in kg.
Body Mass Index (BMI) | 6 weeks
  Body mass index (BMI) is a value derived from the mass (weight) and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
Bone Mass | 6 weeks
  Bone mass means the amount of bone tissue in the skeleton. The bone mass of the patients will be evaluated with the bioelectrical impedance analysis technique. Results will be recorded in kg.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No